CLINICAL TRIAL: NCT05758012
Title: Undesired Effects of Carbetocin Compared To Oxytocin Administered As Single Intravenous Dose or Infusion During Cesarean Delivery: A Prospective Randomised Controlled Study
Brief Title: Carbetocin Compared To Oxytocin During Cesarean Delivery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Collaborators: Ministry of Health, Kuwait (Other Government)
Responsible Party: Principal Investigator, Abdelrady S Ibrahim, MD, Professor of Anesthesia and ICU, Assiut University
Other Study IDs: IRB0000871251
Record Dates: First submitted 2022-11-04; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Cesarean Delivery
MeSH Terms: interventions — Oxytocin; carbetocin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- oxytocin group: Oxytocin 5 IU will be administered by a trained anaesthetist as a one-minute IV injection.
  Interventions: Drug: oxytocin
- Carbetocin group: Carbetocin 100 μg will be administered by a trained anaesthetist as a one-minute IV injection.
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: oxytocin — Participants will be randomized to receive Oxytocin after delivery of the baby's head and shoulders
  Other Names: Syntocinon
  Groups: oxytocin group
Drug: Carbetocin — Participants will be randomized to receive Cabetocin after delivery of the baby's head and shoulders
  Other Names: Pabal
  Groups: Carbetocin group

SUMMARY:
As both oxytocin and carbetocin are used daily in obstetric units all over the world, the investigators find it compelling to investigate whether the hemodynamic and myocardial effects of oxytocin and carbetocin are comparable in healthy women during delivery and determine any potential harmful effects following the use of oxytocin or Carbetocin as uterotonic. Other endpoints relating to uterus tone, blood loss, blood pressure, heart rate, post-operative pain and side effects will also be assessed.

DETAILED DESCRIPTION:
Although the difference between carbetocin and oxytocin in terms of hemodynamic changes, postpartum blood loss and incidence of side effects is not statistically significant. serious cardiovascular adverse events, including ST segment depression, hypotension and tachycardia have been reported after IV oxytocin. Oxytocin dose reduction and/or increased infusion duration may reduce risk of some cardiac-related adverse effects and increase patient safety. As both oxytocin and carbetocin are used daily in obstetric units all over the world, the investigators find it compelling to investigate whether the hemodynamic and myocardial effects of oxytocin and carbetocin are comparable in healthy women during delivery and determine any potential harmful effects following the use of oxytocin or Carbetocin as uterotonic. Other endpoints relating to uterus tone, blood loss, blood pressure, heart rate, post-operative pain and side effects will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Normal singleton pregnancy at gestational age of 36 weeks or more.
* Women with common comorbid diagnoses (diabetes, hypothyroidism, hypertension)
* pregnancy after in vitro fertilization

Exclusion Criteria:

* placenta praevia or invasive placenta.
* pre-eclampsia.
* Bleeding disorder, such as von Willebrand disease type I.
* Current treatment with low-molecular-weight heparin or other anticoagulation medication (not including aspirin).
* Any known intolerance to either of the study drugs.
* Prolonged QT-time.
* Other serious cardiac disease.
* Liver or kidney failure.

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Women will be recruited from the pregnant women attending antenatal clinics in Sabah Maternity Hospital and planned for Delivery either vaginal or Cesarean section .
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Myocardial effects | immediately before drug administration
  Electrocardiograph (QT interval)
Myocardial effects | 24 hours after drug administration
  Electrocardiograph (QT interval)

SECONDARY OUTCOMES:
Cardiac enzyme | immediately before drug administration
  Troponin
Cardiac enzyme | 24 hours after drug administration
  Troponin
Uterine contraction | One hour post delivery
  Palpate the fundus throughout a contraction to determine intensity

CONTACTS AND LOCATIONS:
Overall Officials: Fatemah Qasem, Principal Investigator — Ministry of Health, Kuwait
Locations (1):
- Munistery of Health Kuwait, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: Undecided
the results of the study will be shared with other researchers.

REFERENCES:
- [Background] Masuzawa Y, Kataoka Y, Fujii K, Inoue S. Prophylactic management of postpartum haemorrhage in the third stage of labour: an overview of systematic reviews. Syst Rev. 2018 Oct 11;7(1):156. doi: 10.1186/s13643-018-0817-3. PMID 30305154